CLINICAL TRIAL: NCT06880276
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo Controlled, Parallel Group Study to Assess Efficacy and Safety of QLM3003 Ointment in Participants With Mild or Moderate Atopic Dermatitis
Brief Title: Efficacy and Safety Study of QLM3003 Ointment in Participants With Mild or Moderate Atopic Dermatitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLM3003-301
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1.5% QLM3003 ointment (Experimental): QLM3003 ointment; 1.5%
  Interventions: Drug: 1.5% QLM3003 ointment
- 2% QLM3003 ointment (Experimental): QLM3003 ointment; 2%
  Interventions: Drug: 2% QLM3003 ointment
- Placebo (Placebo Comparator): Vehicle
  Interventions: Drug: QLM3003 Placebo

INTERVENTIONS:
Drug: 1.5% QLM3003 ointment — QLM3003 topical cream; 1.5% cream applied twice daily (BID)
  Arms: 1.5% QLM3003 ointment
Drug: 2% QLM3003 ointment — QLM3003 topical cream; 2% cream applied twice daily (BID)
  Arms: 2% QLM3003 ointment
Drug: QLM3003 Placebo — vehicle; vehicle applied twice daily (BID)
  Arms: Placebo

SUMMARY:
It is a multicenter, randomized, double-blind, placebo-controlled, parallel-group phase 3 clinical trial to evaluate the efficacy of QLM3003 ointment at week 8 based on the primary endpoint (EASI 75) and key secondary endpoint (IGA-TS).in patients with mild to moderate atopic dermatitis. A total of 360 patients with mild to moderate atopic dermatitis are planned to be included and randomized at a ratio of 1:1:1 to receive 1.5% QLM3003 ointment、2% QLM3003 ointment and placebo, twice a day.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-75 years old
* The diagnosis of atopic dermatitis (AD) during screening meets the Hanifin⁃Rajka standard, and the history of AD/ eczema ≥1 year before screening. All of the following conditions must be met during the screening and baseline periods:Number of participants with IGA score of "2" or "3".AD involving the head and neck (scalp excluded), trunk, and extremities, with a total affected BSA of 3-20% (inclusive)

Exclusion Criteria:

* Subjects with comorbidities or other conditions that may interfere with the assessment of the investigational drug or the study disease, as determined by the investigator to be ineligible for participation
* Patients whose current AD disease status was assessed by the investigators to be unstable (spontaneous improvement or rapid deterioration) were not eligible to participate in the study.
* Patients who have received a marketed or investigational biologic for the treatment of AD, such as Dupilumab, within 3 months before baseline or within 5 half-lives of the drug (whichever was longer).
* Patients who had received systemic or topical JAK inhibitor therapy, including but not limited to Tofacitinib, Ruxolitinib, Upadacitinib, Baricitinib, Abrocitinib, Ivarmacitinib, and Gecacitinib, within 4 weeks before baseline or within 5 half-lives of the drug (whichever was longer).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving >=75% Improvement in Eczema Area and Severity Index Total Score (EASI-75) From Baseline at Weeks 8 | Baseline, Week 8
  EASI evaluates severity of participant's AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions(head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in each 4 body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Investigator's Global Assessment (IGA) Score Clear (0) or Almost Clear (1) and a Reduction From Baseline of Greater Than or Equal to ( >=2) Points at Week 8 | Baseline, Week 8
  IGA assesses severity of participant's AD on a 5 point scale. 0= clear, no inflammatory signs of AD; 1= almost clear, AD not fully cleared- light pink residual lesions (except post-inflammatory hyperpigmentation), just perceptible erythema, papulation/induration lichenification, excoriation, and no oozing/crusting; 2= mild AD with light red lesions, slight but definite erythema, papulation/induration, lichenification, excoriation and no oozing/crusting; 3= moderate AD with red lesions, moderate erythema, papulation/induration, lichenification, excoriation and slight oozing/crusting and 4= severe AD with deep dark red lesions, severe erythema, papulation/induration, lichenification, excoriation and moderate to severe oozing/crusting. Higher scores indicating more severity of AD. Assessment excluded soles, palms and scalp.

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Gao, Doctor, Study Director — First Hospital of China Medical University; Furen zhang, Doctor, Study Director — Dermatology Hospital of Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, China